CLINICAL TRIAL: NCT02890537
Title: Treatment of Osteonecrosis of the Femoral Head by Implantation of Preosteoblastic Cells: a Randomized, Controlled, Single Blind Pilot Study
Brief Title: Autologous Osteoblastic Cells Implantation to Early Stage Osteonecrosis of the Femoral Head
Acronym: PREOB-ON2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: University of Liege (Other); Bone Therapeutics S.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2003/281
Record Dates: First submitted 2016-08-25; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Avascular Necrosis of Femur Head
Keywords: Osteonecrosis; Femoral Head; Hip; Orthopedics; Bone; Musculoskeletal Disorders
MeSH Terms: conditions — Femur Head Necrosis; Osteonecrosis; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Core decompression/PREOB® implantation (Experimental): Core decompression/autologous osteoblastic cells (PREOB®) implantation
  Interventions: Drug: Core decompression/PREOB® implantation
- Core decompression/BMC implantation (Active Comparator): Core decompression/bone marrow concentrate (BMC) implantation
  Interventions: Drug: Core decompression/BMC implantation

INTERVENTIONS:
Drug: Core decompression/PREOB® implantation — All subjects received a core decompression under general anesthesia combined with the implantation of PREOB® into the necrotic lesion (single administration).
  Arms: Core decompression/PREOB® implantation
Drug: Core decompression/BMC implantation — All subjects received a core decompression under general anesthesia combined with the implantation of BMC into the necrotic lesion (single administration).
  Arms: Core decompression/BMC implantation

SUMMARY:
Non-traumatic osteonecrosis is a painful disorder of the hip characterized by a necrosis of the osteomedullary tissue, which leads to subchondral bone collapse and joint destruction. Core decompression is currently the treatment of choice for early stage osteonecrosis of the femoral head. This method consists in decompressing the rigid intra-osseous chamber to promote revascularization, thus halting progression of the disease and stimulating repair. Still this treatment remains highly controversial, since the success rates of the first studies have not been repeated.

The exact pathology mechanisms involved in osteonecrosis have not yet be fully elucidated. Several hypotheses have been evoked, including fat embolism, trabecular bone microfractures, microvascular tamponade and, more recently, impaired bone and/or mesenchymal cells recruitment.

Three studies have indicated the potential clinical benefits of cell-based approaches for the treatment of osteonecrosis (Hernigou 1997, Hernigou & Beaujean 2002, Gangji et al. 2004). This is on the basis of these observations that a proprietary population of autologous osteoblastic cells (PREOB®) has been developed.

This Phase 2B study aims at demonstrating the efficacy and safety of PREOB® in the treatment of early stage osteonecrosis of the femoral head. The primary goal of this study was to investigate the safety and efficacy of the implantation of the investigational product PREOB® (human autologous bone marrow-derived osteoblastic cells) in comparison to bone marrow concentrate (BMC) when implanted at the osteonecrotic lesion of the femoral head, with a follow-up period of up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* ARCO stage I or II non-traumatic osteonecrosis of the femoral head, confirmed by conventional X-ray and magnetic resonance imaging (MRI) of the hip
* Aged 18 or higher
* Ability to provide a written, dated and signed informed consent prior to any study-related procedure to understand and comply with study requirements

Exclusion Criteria:

* Evidence of malignant disorder in the past five years
* Positive serology for hepatitis B, hepatitis C, HIV
* Patient unable to undergo a MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2003-10; Primary Completion 2011-05 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of responder subjects | 24 months
  Response defined as the absence of progression to fractural stage (ARCO stage III or higher) & a clinically significant pain improvement
Potential occurrence of any AE or SAE, related to the product or to the procedure, using patient open non-directive questionnaire, physical examination and laboratory measurements | 60 months

SECONDARY OUTCOMES:
Percentage of responder subjects | 3, 6, 12 and 36 months
Percentage of subjects progressing to fractural stage (ARCO stage III or higher), as assessed by conventional X-ray | 3, 6, 12, 24 and 36 months
Change from baseline in VAS pain score | 3, 6, 12, 18, 24, 36 and 48 months
Change from baseline in WOMAC® score | 3, 6, 12, 18, 24, 36 and 48 months
Change from baseline in Lequesne score | 3, 6, 12, 18, 24, 36 and 48 months
Proportion of subjects undergoing a total hip arthroplasty | 6, 12, 24 and 36 months
Time to hip fracture | 36 months

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Investigative site 01, Brussels
  - Investigative site 02, Liège

IPD SHARING:
Plan to Share IPD: No